CLINICAL TRIAL: NCT05159401
Title: The Use of Vibrational Methods of Influencing the Lungs to Restore Their Functional State After Major Reconstructive Cardiac Surgery
Brief Title: The Use of Vibrational Methods of Influencing the Lungs to Restore Their Functional State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Principal Investigator, Aleksandr Eremenko, Clinical Professor, Petrovsky National Research Centre of Surgery
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 09052021
Record Dates: First submitted 2021-11-17; First posted 2021-12-16 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Failure
Keywords: medical rehabilitation; oxygenation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- the first group: the method of vibroacoustic lung massage using the "BARK VibroLUNG" device (Experimental): dynamics blood saturation by pulse oximeter,minute inspiratory lung volume befor/after research
  Interventions: Procedure: prevention of respiratory failure
- the second group:the method of oscillating REР therapy using Acapella DH Green (Experimental): dynamics blood saturation by pulse oximeter,minute inspiratory lung volume befor/after research
  Interventions: Procedure: prevention of respiratory failure
- the third group:the method of hardware stimulation of cough (Comfortable cough Plus) (Experimental): dynamics blood saturation by pulse oximeter,minute inspiratory lung volume befor/after research
  Interventions: Procedure: prevention of respiratory failure
- the fourth group:classical manual chest massage with percussion (Experimental): dynamics blood saturation by pulse oximeter,minute inspiratory lung volume befor/after research
  Interventions: Procedure: prevention of respiratory failure

INTERVENTIONS:
Procedure: prevention of respiratory failure — Positive dynamics during CT or X-ray examinations in the form of reduction of hypoventilation zones, straightening of lung tissue

SUMMARY:
There will be formed of groups for application of vibration methods on the lungs: the method of vibroacoustic lung massage using the "BARK VibroLUNG" device; the method of oscillating PEP therapy using Acapella DH Green; the method of hardware stimulation of cough with a mechanical insufflator-aspirator Comfort Cough Plus (Comfortable cough Plus). As a control group, classical manual chest massage with percussion and verbal stimulation of cough against the background of chest compressions with a total duration of 15 minutes will be used

DETAILED DESCRIPTION:
The patient signs an informed consent to participate in the study after 10-12 hours tracheal extubation and transfer of the patient to spontaneous respiration. The application of one or another method of influence is carried out by the method of random sampling (the envelope method). Next, a session is conducted using one of the methods of vibrational respiratory therapy. We are exploring the gas composition of arterial blood is examined, spirometry, and the respiratory rate is measured after 20 minutes of the procedure. Further, respiratory therapy sessions are repeated 3 times a day for three days

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 years to 80 years inclusive.
2. Performed cardiac surgery in IC conditions.
3. The patient's consent to participate in this study.

Exclusion Criteria:

1. Lack of productive contact with the patient
2. Any disorder in the central nervous system in the perioperative period (acute cerebrovascular accident, coma, posthypoxic encephalopathy), being on a ventilator.
3. Unstable hemodynamics or hemodynamically significant rhythm disturbances
4. Shocks of various etiologies
5. Inability to provide respiratory protection, high risk of aspiration
6. Refusal of the patient to participate in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
the minute inspiratory lung volume | hospitalisation period, an average of 1 week
  Comparison of minute inspiratory lung volume befor/after research using a spirometer
arterial blood oxygenation level | hospitalisation period, an average of 1 day
  Comparison arterial blood oxygenation level before/after researchin the study of arterial blood
SpO2 more than 92% | hospitalisation period, an average of 3 day
  Comparison of SpO2 by pulse oximeter befor/after research (SpO2>92%)

SECONDARY OUTCOMES:
the number of complications | hospitalisation period, an average of 1 week
  Comparison of the number of complications befor/after research
assessment of the duration of hospital stay | hospitalisation period, an average of 1 week
  Comparison of assessment of the duration of hospital stay befor/after research

CONTACTS AND LOCATIONS:
Overall Officials: Alexander А Eremenko, prof, Study Director — Head of the Intensive Care Unit; Darya Ryabova, Principal Investigator — anesthesiologist-resuscitator
Locations (1):
- Petrovsky Research National Center of Surgery, Moscow, Russia

REFERENCES:
- [Derived] Eremenko AA, Zyulyaeva TP, Alferova AP, Fomina DV, Grekova MS, Grin OO, Dmitrieva SS, Molochkov AV, Gens AP, Kotenko KV. [The use of oscillatory respiratory therapy with positive expiratory pressure (PEP-therapy) to restore the functional state of the lungs in patients after cardiac surgery]. Vopr Kurortol Fizioter Lech Fiz Kult. 2023;100(6):21-30. doi: 10.17116/kurort202310006121. Russian. PMID 38289301
- See also: Effectiveness and safety evaluation of a cough stimulation device in early postoperative respiratory rehabilitation in cardiac surgery patients — http://pubmed.ncbi.nlm.nih.gov/34965710/
- See also: Effectiveness of oscillating PEP-therapy in early period after cardiac surgery — http://www.mediasphera.ru/issues/kardiologiya-i-serdechno-sosudistaya-khirurgiya/2021/6/downloads/ru/1199663852021061477
- See also: Comparative Evaluation of Vibratory Physiotherapy Methods in the Early Period after Cardiac Surgery — http://www.vair-journal.com/jour/article/view/603
- See also: Comparing the Inspiratory Capacity Measurements Obtained by Incentive Spirometry and Ultrasonic Spirography in the Early Postoperative Period in Cardiac Surgery Patients — http://www.reanimatology.com/rmt/article/view/2256/1704
- See also: poster report with publication Intensive Care Medicine Experimental. ESICM 2022. 000290 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC9579221/pdf/40635_2022_Article_468.pdf
- See also: poster report with publication Critical Care. 42nd International Symposium on Intensive Care & Emergency Medicine. P330 — http://ccforum.biomedcentral.com/counter/pdf/10.1186/s13054-023-04377-x.pdf